CLINICAL TRIAL: NCT01781923
Title: A Remediation Program for Children at High-Risk of Schizophrenia: 22q11.2 Deletion Syndrome
Brief Title: Cognitive Remediation in 22q11DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Harvard University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00025985; R34MH091314 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: 22q11.2 Deletion Syndrome; Velo-Cardio-Facial Syndrome
Keywords: Cognitive remediation; Social Cognition
MeSH Terms: conditions — DiGeorge Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Remediation (Experimental): 12 week computer-based cognitive remediation program aimed to improve working memory, processing speed, and verbal learning/memory.
  40 week small group social skills training sessions aimed to improve social skills and cognition.
  Interventions: Behavioral: Cognitive remediation program; Behavioral: Small group social skills training
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Cognitive remediation program — Subject plays for 30 minutes, 4 times per week, for 12 weeks.
  Other Names: Posit Science
  Arms: Cognitive Remediation
Behavioral: Small group social skills training — Meet once per week for duration of 40 weeks.
  Arms: Cognitive Remediation

SUMMARY:
The goal of this study is to collect preliminary data on the efficacy of a cognitive remediation program in improving the neurocognitive deficits in children with chromosome 22q11.2 deletion syndrome (22q11DS). This study involves a two part approaching including a computerized cognitive remediation program (CCRP, Posit Science, CA) in combination with a Social Cognitive Training (SCT) program. The computer-based training program has shown encouraging results in improving learning deficits in individuals with schizophrenia and we now seek to adapt them to children with 22q11DS, who have unique needs due to their lower IQ and high risk of psychosis in late adolescence and adulthood. The SCT is a small-group intervention program based on cognitive enhancement therapy, which has been shown to improve social cognition and functionality in adults with schizophrenia. A preliminary study will be performed using this two-pronged approach, to establish the feasibility and gather preliminary data on neurocognition before and after the intervention in these children; these data would enable a larger randomized controlled study to assess the efficacy of this approach.

ELIGIBILITY:
Inclusion Criteria:

* molecular/cytogenetic confirmation of 22q11DS

Exclusion Criteria:

* Intelligence Quotient <60
* diagnosis of psychosis
* pregnancy
* home location does not permit participation in small groups

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in sustained attention | Baseline and 12 weeks
  Sustained attention will be assessed using the Continuous Performance Test.
Change in executive function. | Baseline and 12 weeks
Change in verbal memory. | Baseline and 12 weeks

SECONDARY OUTCOMES:
Social skills | 40 weeks
  Social skills will be measured using a parental survey called the Social Skills Rating System.
Change in brain function and white matter structure. | Baseline and 12 weeks
  The study will examine the impact of CCRP upon brain function and white matter structure in children with 22q11DS.

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Shashi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States